CLINICAL TRIAL: NCT02205736
Title: A Cross Sectional Study of a Breast Health Education Program for Under-served Latino Women in Union and Mecklenburg County
Brief Title: Breast Health Education for Underserved Latino Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: Atrium Health Levine Cancer Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: LCI-BRE-NOS-HEP-001
Record Dates: First submitted 2014-07-29; First posted 2014-07-31 (Estimated); Results first posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-04

CONDITIONS: Breast Cancer
Keywords: Breast health education; Latino women; Group education; Breast cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Living Room Visit participants (Other): Latino women who received breast health education while attending a Living Room Visit.
  Interventions: Other: Breast Health Education

INTERVENTIONS:
Other: Breast Health Education — Small group breast health educational sessions for Latino women in home setting.

SUMMARY:
Subjects will be recruited from the participants in the Union and Mecklenburg County Living Room Visits. Participants in the Living Room Visit will have been recruited using community event flyers. During the Living Room Visits, the Health Educator will provide a general overview of the study. Individuals who are interested in participating in the study will then be generally screened for eligibility by the Protocol Coordinator who will then proceed to provide informed consent to potential subjects.

DETAILED DESCRIPTION:
In an effort to increase early detection of breast cancer our program is designed to remove some of the most common barriers faced by uninsured Latino women including lack of breast health knowledge and inability to pay for screening. The Levine Cancer Institute offers breast cancer education and screening in the growing Latino populations of both Mecklenburg and Union Counties through educational programs known as "Living Room Visits." Living Room Visits are educational sessions hosted at a participant's house that will be led by a Carolinas Healthcare System (CHS) certified bilingual health educator. At least 250 women will participant in the educational sessions between both counties with each session hosting 12-15 participants. Of those women participating in Living Room Visits, those interested will be individually informed of the research opportunity and provided informed consent before being asked to take a pre-test survey. After the educational session, subjects who consented to the study will also complete a post-test survey. Three months after each Living Room Visit, subjects will also be called to complete another post-test survey to assess educational retention. Phone calls and post-test surveys will be administered by Collaborative Institutional Training Initiative (CITI) trained CHS certified bilingual employees only. Analysis of the pre and post-intervention surveys will be administered by a CHS statistician using de-identified data.

ELIGIBILITY:
Inclusion Criteria:

* Latino
* Female
* At least 18 years old
* Resident of Union County or Mecklenburg County, North Carolina

Exclusion Criteria:

* Non-Latino
* Male
* Less than 18 years old
* Not a resident of Union County or Mecklenburg County, North Carolina

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 329 (Actual)
Dates: Start 2014-07; Primary Completion 2016-11 (Actual); Study Completion 2016-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Carrizosa, MD, Principal Investigator — Carolinas Healthcare System, Levine Cancer Institute; Anna Bawtinhimer, BSPH, Study Director — Carolinas Healthcare System, Levine Cancer Institute; Jim Symanowski, PhD, Study Director — Carolinas Healthcare System - Levine Cancer Institute
Locations (1):
- Levine Cancer Institute, Charlotte, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants for the Living Room Visits were recruited by community flyers, word of mouth, and promoted via community gatekeepers.
Groups:
- Living Room Visit Participants: Latino women who received breast health education in community-based small group breast health educational sessions.
Period: Overall Study
Arm/Group | Living Room Visit Participants
Started | 329 (329 participants completed pre- and post-intervention surveys.)
Completed | 223 (223 participants completed the three-month follow-up survey.)
Not Completed | 106
Not completed — Lost to Follow-up | 106

BASELINE CHARACTERISTICS:
Population: 329 participants completed the pre- and post-intervention surveys.
Arm/Group | Living Room Visit Participants
Number analyzed (Participants) | 329
Age, Continuous [Median (Full Range); unit: Years] | 42 [18 to 95]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 329
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 329
  Not Hispanic or Latino | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 329
History of Mammogram (in women aged 40 or older) prior to Living Room Visits [Count of Participants; unit: Participants] — Population: The history of mammogram prior to Living Room Visit will be evaluated in participants aged 40 or older due to current screening recommendations.
  Participants
    number analyzed (Participants) | 195
    (all) | 125

OUTCOME MEASURES:

1. Primary Outcome: The Frequencies of Paired Responses to Identical Questions on a Survey Administered at Two Timepoints: Before the Health Education Program (i.e., Baseline) and Immediately After the Health Education Program (i.e., Post-Intervention).
Description: Participants completed 25-item questionnaires requiring True/False responses to evaluate breast health knowledge at Baseline and Post-Intervention. True/False responses were recoded as being correct or incorrect, resulting in 25 unique 2x2 contingency tables of paired, dichotomous survey responses. Reported here are the frequencies of paired subject responses for each question on the Baseline and Post-Intervention questionnaires.
  Questions are listed below as Row Titles.
  Abbreviations to note include:
  Question: Q Mammography, Mammogram: MAM Breast cancer: BC True/False: T/F
Time Frame: Baseline to Post-Intervention, occurring the same day; duration is approximately several hours.
Population: Latina women, aged 18 years or older at consent (i.e., Baseline), completing both the Baseline and Post-Intervention surveys during the health education program
Measure: Count of Participants; unit: Participants
Groups:
- Living Room Visit Participants: Latina women, aged 18 years or older at consent (i.e., Baseline), completing both the Baseline and Post-Intervention surveys during the Living Room Visits.
Arm/Group | Living Room Visit Participants
Number analyzed (Participants) | 329
Participants
  Q1: MAM is screening that helps doctors look for BC so it can be found early enough to be cured, T/F: Answered incorrectly at Baseline and answered correctly at Post-Intervention | 9
  Q1: MAM is screening that helps doctors look for BC so it can be found early enough to be cured, T/F: Answered incorrectly at Baseline and answered incorrectly at Post-Intervention | 0
  Q1: MAM is screening that helps doctors look for BC so it can be found early enough to be cured, T/F: Answered correctly at Baseline and answered incorrectly at Post-Intervention | 8
  Q1: MAM is screening that helps doctors look for BC so it can be found early enough to be cured, T/F: Answered correctly at Baseline and answered correctly at Post-Intervention | 312
  Q2: MAM is done to stop BC from happening, T/F: Answered incorrectly at Baseline and answered correctly at Post-Intervention | 142
  Q2: MAM is done to stop BC from happening, T/F: Answered incorrectly at Baseline and answered incorrectly at Post-Intervention | 64
  Q2: MAM is done to stop BC from happening, T/F: Answered correctly at Baseline and answered incorrectly at Post-Intervention | 15
  Q2: MAM is done to stop BC from happening, T/F: Answered correctly at Baseline and answered correctly at Post-Intervention | 108
  Q3: MAM does not help to find BC, T/F: Answered incorrectly at Baseline and answered correctly at Post-Intervention | 46
  Q3: MAM does not help to find BC, T/F: Answered incorrectly at Baseline and answered incorrectly at Post-Intervention | 24
  Q3: MAM does not help to find BC, T/F: Answered correctly at Baseline and answered incorrectly at Post-Intervention | 22
  Q3: MAM does not help to find BC, T/F: Answered correctly at Baseline and answered correctly at Post-Intervention | 237
  Q4: Screening MAM are not needed as frequently if you perform regular self-breast exams, T/F: Answered incorrectly at Baseline and answered correctly at Post-Intervention | 36
  Q4: Screening MAM are not needed as frequently if you perform regular self-breast exams, T/F: Answered incorrectly at Baseline and answered incorrectly at Post-Intervention | 11
  Q4: Screening MAM are not needed as frequently if you perform regular self-breast exams, T/F: Answered correctly at Baseline and answered incorrectly at Post-Intervention | 15
  Q4: Screening MAM are not needed as frequently if you perform regular self-breast exams, T/F: Answered correctly at Baseline and answered correctly at Post-Intervention | 267
  Q5: Maintaining a healthy weight may DECREASE your chances of getting BC, T/F: Answered incorrectly at Baseline and answered correctly at Post-Intervention | 143
  Q5: Maintaining a healthy weight may DECREASE your chances of getting BC, T/F: Answered incorrectly at Baseline and answered incorrectly at Post-Intervention | 8
  Q5: Maintaining a healthy weight may DECREASE your chances of getting BC, T/F: Answered correctly at Baseline and answered incorrectly at Post-Intervention | 1
  Q5: Maintaining a healthy weight may DECREASE your chances of getting BC, T/F: Answered correctly at Baseline and answered correctly at Post-Intervention | 177
  Q6: Limiting alcohol intake may DECREASE your chances of getting BC, T/F: Answered incorrectly at Baseline and answered correctly at Post-Intervention | 155
  Q6: Limiting alcohol intake may DECREASE your chances of getting BC, T/F: Answered incorrectly at Baseline and answered incorrectly at Post-Intervention | 8
  Q6: Limiting alcohol intake may DECREASE your chances of getting BC, T/F: Answered correctly at Baseline and answered incorrectly at Post-Intervention | 4
  Q6: Limiting alcohol intake may DECREASE your chances of getting BC, T/F: Answered correctly at Baseline and answered correctly at Post-Intervention | 162
  Q7: Regular physical activity/exercise may DECREASE your chances of getting BC, T/F: Answered incorrectly at Baseline and answered correctly at Post-Intervention | 113
  Q7: Regular physical activity/exercise may DECREASE your chances of getting BC, T/F: Answered incorrectly at Baseline and answered incorrectly at Post-Intervention | 4
  Q7: Regular physical activity/exercise may DECREASE your chances of getting BC, T/F: Answered correctly at Baseline and answered incorrectly at Post-Intervention | 0
  Q7: Regular physical activity/exercise may DECREASE your chances of getting BC, T/F: Answered correctly at Baseline and answered correctly at Post-Intervention | 212
  Q8: Breastfeeding may DECREASE your chances of getting BC, T/F: Answered incorrectly at Baseline and answered correctly at Post-Intervention | 109
  Q8: Breastfeeding may DECREASE your chances of getting BC, T/F: Answered incorrectly at Baseline and answered incorrectly at Post-Intervention | 13
  Q8: Breastfeeding may DECREASE your chances of getting BC, T/F: Answered correctly at Baseline and answered incorrectly at Post-Intervention | 4
  Q8: Breastfeeding may DECREASE your chances of getting BC, T/F: Answered correctly at Baseline and answered correctly at Post-Intervention | 203
  Q9: Having large breasts may INCREASE your chances of getting BC, T/F: Answered incorrectly at Baseline and answered correctly at Post-Intervention | 39
  Q9: Having large breasts may INCREASE your chances of getting BC, T/F: Answered incorrectly at Baseline and answered incorrectly at Post-Intervention | 5
  Q9: Having large breasts may INCREASE your chances of getting BC, T/F: Answered correctly at Baseline and answered incorrectly at Post-Intervention | 4
  Q9: Having large breasts may INCREASE your chances of getting BC, T/F: Answered correctly at Baseline and answered correctly at Post-Intervention | 281
  Q10: Trauma or injury to the breast(s) may INCREASE your chances of getting BC, T/F: Answered incorrectly at Baseline and answered correctly at Post-Intervention | 219
  Q10: Trauma or injury to the breast(s) may INCREASE your chances of getting BC, T/F: Answered incorrectly at Baseline and answered incorrectly at Post-Intervention | 16
  Q10: Trauma or injury to the breast(s) may INCREASE your chances of getting BC, T/F: Answered correctly at Baseline and answered incorrectly at Post-Intervention | 4
  Q10: Trauma or injury to the breast(s) may INCREASE your chances of getting BC, T/F: Answered correctly at Baseline and answered correctly at Post-Intervention | 90
  Q11: Having a mother with BC may INCREASE your chances of getting BC, T/F: Answered incorrectly at Baseline and answered correctly at Post-Intervention | 25
  Q11: Having a mother with BC may INCREASE your chances of getting BC, T/F: Answered incorrectly at Baseline and answered incorrectly at Post-Intervention | 2
  Q11: Having a mother with BC may INCREASE your chances of getting BC, T/F: Answered correctly at Baseline and answered incorrectly at Post-Intervention | 2
  Q11: Having a mother with BC may INCREASE your chances of getting BC, T/F: Answered correctly at Baseline and answered correctly at Post-Intervention | 300
  Q12: Having a friend with BC may INCREASE your chances of getting BC, T/F: Answered incorrectly at Baseline and answered correctly at Post-Intervention | 13
  Q12: Having a friend with BC may INCREASE your chances of getting BC, T/F: Answered incorrectly at Baseline and answered incorrectly at Post-Intervention | 0
  Q12: Having a friend with BC may INCREASE your chances of getting BC, T/F: Answered correctly at Baseline and answered incorrectly at Post-Intervention | 3
  Q12: Having a friend with BC may INCREASE your chances of getting BC, T/F: Answered correctly at Baseline and answered correctly at Post-Intervention | 313
  Q13: Having an aunt with B/C may INCREASE your chances of getting B/C, T/F: Answered incorrectly at Baseline and answered correctly at Post-Intervention | 76
  Q13: Having an aunt with B/C may INCREASE your chances of getting B/C, T/F: Answered incorrectly at Baseline and answered incorrectly at Post-Intervention | 4
  Q13: Having an aunt with B/C may INCREASE your chances of getting B/C, T/F: Answered correctly at Baseline and answered incorrectly at Post-Intervention | 2
  Q13: Having an aunt with B/C may INCREASE your chances of getting B/C, T/F: Answered correctly at Baseline and answered correctly at Post-Intervention | 247
  Q14: You should go see a doctor if you notice changes in the size or shape of your breast(s), T/F: Answered incorrectly at Baseline and answered correctly at Post-Intervention | 6
  Q14: You should go see a doctor if you notice changes in the size or shape of your breast(s), T/F: Answered incorrectly at Baseline and answered incorrectly at Post-Intervention | 0
  Q14: You should go see a doctor if you notice changes in the size or shape of your breast(s), T/F: Answered correctly at Baseline and answered incorrectly at Post-Intervention | 1
  Q14: You should go see a doctor if you notice changes in the size or shape of your breast(s), T/F: Answered correctly at Baseline and answered correctly at Post-Intervention | 322
  Q15: See a doctor if you find unusual liquid coming from nipple when not pregnant/breastfeeding, T/F: Answered incorrectly at Baseline and answered correctly at Post-Intervention | 6
  Q15: See a doctor if you find unusual liquid coming from nipple when not pregnant/breastfeeding, T/F: Answered incorrectly at Baseline and answered incorrectly at Post-Intervention | 1
  Q15: See a doctor if you find unusual liquid coming from nipple when not pregnant/breastfeeding, T/F: Answered correctly at Baseline and answered incorrectly at Post-Intervention | 0
  Q15: See a doctor if you find unusual liquid coming from nipple when not pregnant/breastfeeding, T/F: Answered correctly at Baseline and answered correctly at Post-Intervention | 322
  Q16: See a doctor if you have a stabbing breast pain that does not seem to get better, T/F: Answered incorrectly at Baseline and answered correctly at Post-Intervention | 5
  Q16: See a doctor if you have a stabbing breast pain that does not seem to get better, T/F: Answered incorrectly at Baseline and answered incorrectly at Post-Intervention | 0
  Q16: See a doctor if you have a stabbing breast pain that does not seem to get better, T/F: Answered correctly at Baseline and answered incorrectly at Post-Intervention | 1
  Q16: See a doctor if you have a stabbing breast pain that does not seem to get better, T/F: Answered correctly at Baseline and answered correctly at Post-Intervention | 323
  Q17: See a doctor if you notice pulling in of the nipple or other parts of your breast(s), T/F: Answered incorrectly at Baseline and answered correctly at Post-Intervention | 16
  Q17: See a doctor if you notice pulling in of the nipple or other parts of your breast(s), T/F: Answered incorrectly at Baseline and answered incorrectly at Post-Intervention | 0
  Q17: See a doctor if you notice pulling in of the nipple or other parts of your breast(s), T/F: Answered correctly at Baseline and answered incorrectly at Post-Intervention | 0
  Q17: See a doctor if you notice pulling in of the nipple or other parts of your breast(s), T/F: Answered correctly at Baseline and answered correctly at Post-Intervention | 313
  Q18: Women don't need to be aware of changes with their breasts until they reach 40 years old, T/F: Answered incorrectly at Baseline and answered correctly at Post-Intervention | 25
  Q18: Women don't need to be aware of changes with their breasts until they reach 40 years old, T/F: Answered incorrectly at Baseline and answered incorrectly at Post-Intervention | 15
  Q18: Women don't need to be aware of changes with their breasts until they reach 40 years old, T/F: Answered correctly at Baseline and answered incorrectly at Post-Intervention | 15
  Q18: Women don't need to be aware of changes with their breasts until they reach 40 years old, T/F: Answered correctly at Baseline and answered correctly at Post-Intervention | 274
  Q19: Knowing how your breast/underarms normally look/feel are important parts of breast health, T/F: Answered incorrectly at Baseline and answered correctly at Post-Intervention | 18
  Q19: Knowing how your breast/underarms normally look/feel are important parts of breast health, T/F: Answered incorrectly at Baseline and answered incorrectly at Post-Intervention | 1
  Q19: Knowing how your breast/underarms normally look/feel are important parts of breast health, T/F: Answered correctly at Baseline and answered incorrectly at Post-Intervention | 3
  Q19: Knowing how your breast/underarms normally look/feel are important parts of breast health, T/F: Answered correctly at Baseline and answered correctly at Post-Intervention | 307
  Q20: A screening MAM is only needed if you noticed changes with your breast(s) in the past year, T/F: Answered incorrectly at Baseline and answered correctly at Post-Intervention | 62
  Q20: A screening MAM is only needed if you noticed changes with your breast(s) in the past year, T/F: Answered incorrectly at Baseline and answered incorrectly at Post-Intervention | 17
  Q20: A screening MAM is only needed if you noticed changes with your breast(s) in the past year, T/F: Answered correctly at Baseline and answered incorrectly at Post-Intervention | 13
  Q20: A screening MAM is only needed if you noticed changes with your breast(s) in the past year, T/F: Answered correctly at Baseline and answered correctly at Post-Intervention | 237
  Q21: When detected early, the chance of curing breast cancer is increased, T/F: Answered incorrectly at Baseline and answered correctly at Post-Intervention | 3
  Q21: When detected early, the chance of curing breast cancer is increased, T/F: Answered incorrectly at Baseline and answered incorrectly at Post-Intervention | 0
  Q21: When detected early, the chance of curing breast cancer is increased, T/F: Answered correctly at Baseline and answered incorrectly at Post-Intervention | 10
  Q21: When detected early, the chance of curing breast cancer is increased, T/F: Answered correctly at Baseline and answered correctly at Post-Intervention | 316
  Q22: Getting yearly MAM and clinical breast exams are the best ways to detect BC early, T/F: Answered incorrectly at Baseline and answered correctly at Post-Intervention | 9
  Q22: Getting yearly MAM and clinical breast exams are the best ways to detect BC early, T/F: Answered incorrectly at Baseline and answered incorrectly at Post-Intervention | 4
  Q22: Getting yearly MAM and clinical breast exams are the best ways to detect BC early, T/F: Answered correctly at Baseline and answered incorrectly at Post-Intervention | 10
  Q22: Getting yearly MAM and clinical breast exams are the best ways to detect BC early, T/F: Answered correctly at Baseline and answered correctly at Post-Intervention | 306
  Q23: BC is the most common cancer diagnosed among Hispanic/Latina women, T/F: Answered incorrectly at Baseline and answered correctly at Post-Intervention | 75
  Q23: BC is the most common cancer diagnosed among Hispanic/Latina women, T/F: Answered incorrectly at Baseline and answered incorrectly at Post-Intervention | 7
  Q23: BC is the most common cancer diagnosed among Hispanic/Latina women, T/F: Answered correctly at Baseline and answered incorrectly at Post-Intervention | 8
  Q23: BC is the most common cancer diagnosed among Hispanic/Latina women, T/F: Answered correctly at Baseline and answered correctly at Post-Intervention | 239
  Q24: Healthy women do not need to get MAM annually, T/F: Answered incorrectly at Baseline and answered correctly at Post-Intervention | 31
  Q24: Healthy women do not need to get MAM annually, T/F: Answered incorrectly at Baseline and answered incorrectly at Post-Intervention | 8
  Q24: Healthy women do not need to get MAM annually, T/F: Answered correctly at Baseline and answered incorrectly at Post-Intervention | 9
  Q24: Healthy women do not need to get MAM annually, T/F: Answered correctly at Baseline and answered correctly at Post-Intervention | 281
  Q25: If you don't see changes with your breasts in the past year, a MAM isn't necessary, T/F: Answered incorrectly at Baseline and answered correctly at Post-Intervention | 49
  Q25: If you don't see changes with your breasts in the past year, a MAM isn't necessary, T/F: Answered incorrectly at Baseline and answered incorrectly at Post-Intervention | 13
  Q25: If you don't see changes with your breasts in the past year, a MAM isn't necessary, T/F: Answered correctly at Baseline and answered incorrectly at Post-Intervention | 7
  Q25: If you don't see changes with your breasts in the past year, a MAM isn't necessary, T/F: Answered correctly at Baseline and answered correctly at Post-Intervention | 260
Statistical Analysis 1: Comparison: Living Room Visit Participants; Patients gave True/False responses to Question 1 at Baseline and Post-Intervention; the True/False responses were mapped to being correct or incorrect. The null hypothesis was that the intervention had no effect on breast health, or that the probability of answering incorrectly on the Baseline questionnaire and correctly on the Post-Intervention questionnaire was equal to the probability of answering correctly on the Baseline questionnaire and incorrectly on the Post-Intervention questionnaire; Test type: Superiority; p = 0.8084, McNemar — Each of the 25 co-primary objectives were tested at the 2-sided, Bonferroni-corrected alpha=0.002 significance level to preserve an overall type I error rate of 5%
Statistical Analysis 2: Comparison: Living Room Visit Participants; Patients gave True/False responses to Question 2 at Baseline and Post-Intervention; the True/False responses were mapped to being correct or incorrect. The null hypothesis was that the intervention had no effect on breast health, or that the probability of answering incorrectly on the Baseline questionnaire and correctly on the Post-Intervention questionnaire was equal to the probability of answering correctly on the Baseline questionnaire and incorrectly on the Post-Intervention questionnaire; Test type: Superiority; p < .0001, McNemar — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Living Room Visit Participants; Patients gave True/False responses to Question 3 at Baseline and Post-Intervention; the True/False responses were mapped to being correct or incorrect. The null hypothesis was that the intervention had no effect on breast health, or that the probability of answering incorrectly on the Baseline questionnaire and correctly on the Post-Intervention questionnaire was equal to the probability of answering correctly on the Baseline questionnaire and incorrectly on the Post-Intervention questionnaire; Test type: Superiority; p = 0.0036, McNemar — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 4: Comparison: Living Room Visit Participants; Patients gave True/False responses to Question 4 at Baseline and Post-Intervention; the True/False responses were mapped to being correct or incorrect. The null hypothesis was that the intervention had no effect on breast health, or that the probability of answering incorrectly on the Baseline questionnaire and correctly on the Post-Intervention questionnaire was equal to the probability of answering correctly on the Baseline questionnaire and incorrectly on the Post-Intervention questionnaire; Test type: Superiority; p = 0.0033, McNemar — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 5: Comparison: Living Room Visit Participants; Patients gave True/False responses to Question 5 at Baseline and Post-Intervention; the True/False responses were mapped to being correct or incorrect. The null hypothesis was that the intervention had no effect on breast health, or that the probability of answering incorrectly on the Baseline questionnaire and correctly on the Post-Intervention questionnaire was equal to the probability of answering correctly on the Baseline questionnaire and incorrectly on the Post-Intervention questionnaire; Test type: Superiority; p < .0001, McNemar — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 6: Comparison: Living Room Visit Participants; Patients gave True/False responses to Question 6 at Baseline and Post-Intervention; the True/False responses were mapped to being correct or incorrect. The null hypothesis was that the intervention had no effect on breast health, or that the probability of answering incorrectly on the Baseline questionnaire and correctly on the Post-Intervention questionnaire was equal to the probability of answering correctly on the Baseline questionnaire and incorrectly on the Post-Intervention questionnaire; Test type: Superiority; p < .0001, McNemar — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 7: Comparison: Living Room Visit Participants; Patients gave True/False responses to Question 7 at Baseline and Post-Intervention; the True/False responses were mapped to being correct or incorrect. The null hypothesis was that the intervention had no effect on breast health, or that the probability of answering incorrectly on the Baseline questionnaire and correctly on the Post-Intervention questionnaire was equal to the probability of answering correctly on the Baseline questionnaire and incorrectly on the Post-Intervention questionnaire; Test type: Superiority; p < .0001, McNemar — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 8: Comparison: Living Room Visit Participants; Patients gave True/False responses to Question 8 at Baseline and Post-Intervention; the True/False responses were mapped to being correct or incorrect. The null hypothesis was that the intervention had no effect on breast health, or that the probability of answering incorrectly on the Baseline questionnaire and correctly on the Post-Intervention questionnaire was equal to the probability of answering correctly on the Baseline questionnaire and incorrectly on the Post-Intervention questionnaire; Test type: Superiority; p < .0001, McNemar — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 9: Comparison: Living Room Visit Participants; Patients gave True/False responses to Question 9 at Baseline and Post-Intervention; the True/False responses were mapped to being correct or incorrect. The null hypothesis was that the intervention had no effect on breast health, or that the probability of answering incorrectly on the Baseline questionnaire and correctly on the Post-Intervention questionnaire was equal to the probability of answering correctly on the Baseline questionnaire and incorrectly on the Post-Intervention questionnaire; Test type: Superiority; p < .0001, McNemar — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 10: Comparison: Living Room Visit Participants; Patients gave True/False responses to Question 10 at Baseline and Post-Intervention; the True/False responses were mapped to being correct or incorrect. The null hypothesis was that the intervention had no effect on breast health, or that the probability of answering incorrectly on the Baseline questionnaire and correctly on the Post-Intervention questionnaire was equal to the probability of answering correctly on the Baseline questionnaire and incorrectly on the Post-Intervention questionnaire; Test type: Superiority; p < .0001, McNemar — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 11: Comparison: Living Room Visit Participants; Patients gave True/False responses to Question 11 at Baseline and Post-Intervention; the True/False responses were mapped to being correct or incorrect. The null hypothesis was that the intervention had no effect on breast health, or that the probability of answering incorrectly on the Baseline questionnaire and correctly on the Post-Intervention questionnaire was equal to the probability of answering correctly on the Baseline questionnaire and incorrectly on the Post-Intervention questionnaire; Test type: Superiority; p < .0001, McNemar — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 12: Comparison: Living Room Visit Participants; Patients gave True/False responses to Question 12 at Baseline and Post-Intervention; the True/False responses were mapped to being correct or incorrect. The null hypothesis was that the intervention had no effect on breast health, or that the probability of answering incorrectly on the Baseline questionnaire and correctly on the Post-Intervention questionnaire was equal to the probability of answering correctly on the Baseline questionnaire and incorrectly on the Post-Intervention questionnaire; Test type: Superiority; p = 0.0124, McNemar — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 13: Comparison: Living Room Visit Participants; Patients gave True/False responses to Question 13 at Baseline and Post-Intervention; the True/False responses were mapped to being correct or incorrect. The null hypothesis was that the intervention had no effect on breast health, or that the probability of answering incorrectly on the Baseline questionnaire and correctly on the Post-Intervention questionnaire was equal to the probability of answering correctly on the Baseline questionnaire and incorrectly on the Post-Intervention questionnaire; Test type: Superiority; p < .0001, McNemar — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 14: Comparison: Living Room Visit Participants; Patients gave True/False responses to Question 14 at Baseline and Post-Intervention; the True/False responses were mapped to being correct or incorrect. The null hypothesis was that the intervention had no effect on breast health, or that the probability of answering incorrectly on the Baseline questionnaire and correctly on the Post-Intervention questionnaire was equal to the probability of answering correctly on the Baseline questionnaire and incorrectly on the Post-Intervention questionnaire; Test type: Superiority; p = 0.0588, McNemar — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 15: Comparison: Living Room Visit Participants; Patients gave True/False responses to Question 15 at Baseline and Post-Intervention; the True/False responses were mapped to being correct or incorrect. The null hypothesis was that the intervention had no effect on breast health, or that the probability of answering incorrectly on the Baseline questionnaire and correctly on the Post-Intervention questionnaire was equal to the probability of answering correctly on the Baseline questionnaire and incorrectly on the Post-Intervention questionnaire; Test type: Superiority; p = 0.0143, McNemar — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 16: Comparison: Living Room Visit Participants; Patients gave True/False responses to Question 16 at Baseline and Post-Intervention; the True/False responses were mapped to being correct or incorrect. The null hypothesis was that the intervention had no effect on breast health, or that the probability of answering incorrectly on the Baseline questionnaire and correctly on the Post-Intervention questionnaire was equal to the probability of answering correctly on the Baseline questionnaire and incorrectly on the Post-Intervention questionnaire; Test type: Superiority; p = 0.1025, McNemar — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 17: Comparison: Living Room Visit Participants; Patients gave True/False responses to Question 17 at Baseline and Post-Intervention; the True/False responses were mapped to being correct or incorrect. The null hypothesis was that the intervention had no effect on breast health, or that the probability of answering incorrectly on the Baseline questionnaire and correctly on the Post-Intervention questionnaire was equal to the probability of answering correctly on the Baseline questionnaire and incorrectly on the Post-Intervention questionnaire; Test type: Superiority; p = 0.0001, McNemar — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 18: Comparison: Living Room Visit Participants; Patients gave True/False responses to Question 18 at Baseline and Post-Intervention; the True/False responses were mapped to being correct or incorrect. The null hypothesis was that the intervention had no effect on breast health, or that the probability of answering incorrectly on the Baseline questionnaire and correctly on the Post-Intervention questionnaire was equal to the probability of answering correctly on the Baseline questionnaire and incorrectly on the Post-Intervention questionnaire; Test type: Superiority; p = 0.1138, McNemar — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 19: Comparison: Living Room Visit Participants; Patients gave True/False responses to Question 19 at Baseline and Post-Intervention; the True/False responses were mapped to being correct or incorrect. The null hypothesis was that the intervention had no effect on breast health, or that the probability of answering incorrectly on the Baseline questionnaire and correctly on the Post-Intervention questionnaire was equal to the probability of answering correctly on the Baseline questionnaire and incorrectly on the Post-Intervention questionnaire; Test type: Superiority; p = 0.0011, McNemar — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 20: Comparison: Living Room Visit Participants; Patients gave True/False responses to Question 20 at Baseline and Post-Intervention; the True/False responses were mapped to being correct or incorrect. The null hypothesis was that the intervention had no effect on breast health, or that the probability of answering incorrectly on the Baseline questionnaire and correctly on the Post-Intervention questionnaire was equal to the probability of answering correctly on the Baseline questionnaire and incorrectly on the Post-Intervention questionnaire; Test type: Superiority; p < .0001, McNemar — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 21: Comparison: Living Room Visit Participants; Patients gave True/False responses to Question 21 at Baseline and Post-Intervention; the True/False responses were mapped to being correct or incorrect. The null hypothesis was that the intervention had no effect on breast health, or that the probability of answering incorrectly on the Baseline questionnaire and correctly on the Post-Intervention questionnaire was equal to the probability of answering correctly on the Baseline questionnaire and incorrectly on the Post-Intervention questionnaire; Test type: Superiority; p = 0.0522, McNemar — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 22: Comparison: Living Room Visit Participants; Patients gave True/False responses to Question 22 at Baseline and Post-Intervention; the True/False responses were mapped to being correct or incorrect. The null hypothesis was that the intervention had no effect on breast health, or that the probability of answering incorrectly on the Baseline questionnaire and correctly on the Post-Intervention questionnaire was equal to the probability of answering correctly on the Baseline questionnaire and incorrectly on the Post-Intervention questionnaire; Test type: Superiority; p = 0.8185, McNemar — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 23: Comparison: Living Room Visit Participants; Patients gave True/False responses to Question 24 at Baseline and Post-Intervention; the True/False responses were mapped to being correct or incorrect. The null hypothesis was that the intervention had no effect on breast health, or that the probability of answering incorrectly on the Baseline questionnaire and correctly on the Post-Intervention questionnaire was equal to the probability of answering correctly on the Baseline questionnaire and incorrectly on the Post-Intervention questionnaire; Test type: Superiority; p = 0.0005, McNemar — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 24: Comparison: Living Room Visit Participants; Subjects recorded True/False answers to Q25 at Baseline and Post-Intervention; the True/False responses were mapped to being correct or incorrect. The contingency table of 329 responses to Q25 displayed the following: N=260 Correct at Baseline and Correct at Post-Intervention (79.0%), N=7 Correct at Baseline and Incorrect at Post-Intervention (2.1%), N=49 Incorrect at Baseline and Correct at Post-Intervention (14.9%), N=13 Incorrect at Baseline and Incorrect at Post-Intervention (4.0%); Test type: Superiority; p < .0001, McNemar — [p-value comment as in outcome 1, analysis 1]

2. Secondary Outcome: The Frequencies of Paired Responses to Identical Questions on a Survey Administered at Two Timepoints: Before the Health Education Program (i.e., Baseline) and Three Months After the Intervention to Assess Retention (i.e., 3-Month Contact)
Description: Participants completed 25-item questionnaires requiring True/False responses to evaluate breast health knowledge at Baseline and 3-Month Contact. True/False responses were recoded as being correct or incorrect, resulting in 25 unique 2x2 contingency tables of paired, dichotomous survey responses. Reported here are the frequencies of paired subject responses for each question on the Baseline and 3-Month Contact questionnaires.
  Questions are listed below as Row Titles.
  Abbreviations to note include:
  Question: Q Mammography, Mammogram: MAM Breast cancer: BC True/False: T/F
Time Frame: Baseline to 3-Month Contact; duration is approximately three months
Population: Latina women, aged 18 years or older at consent (i.e., baseline), completing both the Baseline and 3-month Contact surveys following the breast health education program. This outcome is reported only for subjects completing the 3-month Contact survey.
Measure: Count of Participants; unit: Participants
Groups:
- Living Room Visit Participants: Latina women, aged 18 years or older at consent (i.e., baseline), completing both the Baseline and 3-month Contact surveys during the Living Room Visits (i.e., breast health education program).
Arm/Group | Living Room Visit Participants
Number analyzed (Participants) | 223
Participants
  Q1: MAM is screening that helps doctors look for BC so it can be found early enough to be cured, T/F: Answered incorrectly at Baseline and answered correctly at 3-Month Contact | 8
  Q1: MAM is screening that helps doctors look for BC so it can be found early enough to be cured, T/F: Answered incorrectly at Baseline and answered incorrectly at 3-Month Contact | 0
  Q1: MAM is screening that helps doctors look for BC so it can be found early enough to be cured, T/F: Answered correctly at Baseline and answered incorrectly at 3-Month Contact | 4
  Q1: MAM is screening that helps doctors look for BC so it can be found early enough to be cured, T/F: Answered correctly at Baseline and answered correctly at 3-Month Contact | 211
  Q2: MAM is done to stop BC from happening, T/F: Answered incorrectly at Baseline and answered correctly at 3-Month Contact | 68
  Q2: MAM is done to stop BC from happening, T/F: Answered incorrectly at Baseline and answered incorrectly at 3-Month Contact | 74
  Q2: MAM is done to stop BC from happening, T/F: Answered correctly at Baseline and answered incorrectly at 3-Month Contact | 15
  Q2: MAM is done to stop BC from happening, T/F: Answered correctly at Baseline and answered correctly at 3-Month Contact | 66
  Q3: MAM does not help to find BC, T/F: Answered incorrectly at Baseline and answered correctly at 3-Month Contact | 45
  Q3: MAM does not help to find BC, T/F: Answered incorrectly at Baseline and answered incorrectly at 3-Month Contact | 7
  Q3: MAM does not help to find BC, T/F: Answered correctly at Baseline and answered incorrectly at 3-Month Contact | 22
  Q3: MAM does not help to find BC, T/F: Answered correctly at Baseline and answered correctly at 3-Month Contact | 149
  Q4: Screening MAM are not needed as frequently if you perform regular self-breast exams, T/F: Answered incorrectly at Baseline and answered correctly at 3-Month Contact | 27
  Q4: Screening MAM are not needed as frequently if you perform regular self-breast exams, T/F: Answered incorrectly at Baseline and answered incorrectly at 3-Month Contact | 8
  Q4: Screening MAM are not needed as frequently if you perform regular self-breast exams, T/F: Answered correctly at Baseline and answered incorrectly at 3-Month Contact | 14
  Q4: Screening MAM are not needed as frequently if you perform regular self-breast exams, T/F: Answered correctly at Baseline and answered correctly at 3-Month Contact | 174
  Q5: Maintaining a healthy weight may DECREASE your chances of getting BC, T/F: Answered incorrectly at Baseline and answered correctly at 3-Month Contact | 75
  Q5: Maintaining a healthy weight may DECREASE your chances of getting BC, T/F: Answered incorrectly at Baseline and answered incorrectly at 3-Month Contact | 28
  Q5: Maintaining a healthy weight may DECREASE your chances of getting BC, T/F: Answered correctly at Baseline and answered incorrectly at 3-Month Contact | 18
  Q5: Maintaining a healthy weight may DECREASE your chances of getting BC, T/F: Answered correctly at Baseline and answered correctly at 3-Month Contact | 102
  Q6: Limiting alcohol intake may DECREASE your chances of getting BC, T/F: Answered incorrectly at Baseline and answered correctly at 3-Month Contact | 72
  Q6: Limiting alcohol intake may DECREASE your chances of getting BC, T/F: Answered incorrectly at Baseline and answered incorrectly at 3-Month Contact | 42
  Q6: Limiting alcohol intake may DECREASE your chances of getting BC, T/F: Answered correctly at Baseline and answered incorrectly at 3-Month Contact | 15
  Q6: Limiting alcohol intake may DECREASE your chances of getting BC, T/F: Answered correctly at Baseline and answered correctly at 3-Month Contact | 94
  Q7: Regular physical activity/exercise may DECREASE your chances of getting BC, T/F: Answered incorrectly at Baseline and answered correctly at 3-Month Contact | 62
  Q7: Regular physical activity/exercise may DECREASE your chances of getting BC, T/F: Answered incorrectly at Baseline and answered incorrectly at 3-Month Contact | 20
  Q7: Regular physical activity/exercise may DECREASE your chances of getting BC, T/F: Answered correctly at Baseline and answered incorrectly at 3-Month Contact | 18
  Q7: Regular physical activity/exercise may DECREASE your chances of getting BC, T/F: Answered correctly at Baseline and answered correctly at 3-Month Contact | 123
  Q8: Breastfeeding may DECREASE your chances of getting BC, T/F: Answered incorrectly at Baseline and answered correctly at 3-Month Contact | 44
  Q8: Breastfeeding may DECREASE your chances of getting BC, T/F: Answered incorrectly at Baseline and answered incorrectly at 3-Month Contact | 41
  Q8: Breastfeeding may DECREASE your chances of getting BC, T/F: Answered correctly at Baseline and answered incorrectly at 3-Month Contact | 15
  Q8: Breastfeeding may DECREASE your chances of getting BC, T/F: Answered correctly at Baseline and answered correctly at 3-Month Contact | 123
  Q9: Having large breasts may INCREASE your chances of getting BC, T/F: Answered incorrectly at Baseline and answered correctly at 3-Month Contact | 18
  Q9: Having large breasts may INCREASE your chances of getting BC, T/F: Answered incorrectly at Baseline and answered incorrectly at 3-Month Contact | 13
  Q9: Having large breasts may INCREASE your chances of getting BC, T/F: Answered correctly at Baseline and answered incorrectly at 3-Month Contact | 20
  Q9: Having large breasts may INCREASE your chances of getting BC, T/F: Answered correctly at Baseline and answered correctly at 3-Month Contact | 172
  Q10: Trauma or injury to the breast(s) may INCREASE your chances of getting BC, T/F: Answered incorrectly at Baseline and answered correctly at 3-Month Contact | 94
  Q10: Trauma or injury to the breast(s) may INCREASE your chances of getting BC, T/F: Answered incorrectly at Baseline and answered incorrectly at 3-Month Contact | 71
  Q10: Trauma or injury to the breast(s) may INCREASE your chances of getting BC, T/F: Answered correctly at Baseline and answered incorrectly at 3-Month Contact | 11
  Q10: Trauma or injury to the breast(s) may INCREASE your chances of getting BC, T/F: Answered correctly at Baseline and answered correctly at 3-Month Contact | 47
  Q11: Having a mother with BC may INCREASE your chances of getting BC, T/F: Answered incorrectly at Baseline and answered correctly at 3-Month Contact | 18
  Q11: Having a mother with BC may INCREASE your chances of getting BC, T/F: Answered incorrectly at Baseline and answered incorrectly at 3-Month Contact | 4
  Q11: Having a mother with BC may INCREASE your chances of getting BC, T/F: Answered correctly at Baseline and answered incorrectly at 3-Month Contact | 4
  Q11: Having a mother with BC may INCREASE your chances of getting BC, T/F: Answered correctly at Baseline and answered correctly at 3-Month Contact | 197
  Q12: Having a friend with BC may INCREASE your chances of getting BC, T/F: Answered incorrectly at Baseline and answered correctly at 3-Month Contact | 11
  Q12: Having a friend with BC may INCREASE your chances of getting BC, T/F: Answered incorrectly at Baseline and answered incorrectly at 3-Month Contact | 0
  Q12: Having a friend with BC may INCREASE your chances of getting BC, T/F: Answered correctly at Baseline and answered incorrectly at 3-Month Contact | 4
  Q12: Having a friend with BC may INCREASE your chances of getting BC, T/F: Answered correctly at Baseline and answered correctly at 3-Month Contact | 208
  Q13: Having an aunt with B/C may INCREASE your chances of getting B/C, T/F: Answered incorrectly at Baseline and answered correctly at 3-Month Contact | 32
  Q13: Having an aunt with B/C may INCREASE your chances of getting B/C, T/F: Answered incorrectly at Baseline and answered incorrectly at 3-Month Contact | 20
  Q13: Having an aunt with B/C may INCREASE your chances of getting B/C, T/F: Answered correctly at Baseline and answered incorrectly at 3-Month Contact | 12
  Q13: Having an aunt with B/C may INCREASE your chances of getting B/C, T/F: Answered correctly at Baseline and answered correctly at 3-Month Contact | 159
  Q14: You should go see a doctor if you notice changes in the size or shape of your breast(s), T/F: Answered incorrectly at Baseline and answered correctly at 3-Month Contact | 4
  Q14: You should go see a doctor if you notice changes in the size or shape of your breast(s), T/F: Answered incorrectly at Baseline and answered incorrectly at 3-Month Contact | 0
  Q14: You should go see a doctor if you notice changes in the size or shape of your breast(s), T/F: Answered correctly at Baseline and answered incorrectly at 3-Month Contact | 1
  Q14: You should go see a doctor if you notice changes in the size or shape of your breast(s), T/F: Answered correctly at Baseline and answered correctly at 3-Month Contact | 218
  Q15: See a doctor if you find unusual liquid coming from nipple when not pregnant/breastfeeding, T/F: Answered incorrectly at Baseline and answered correctly at 3-Month Contact | 3
  Q15: See a doctor if you find unusual liquid coming from nipple when not pregnant/breastfeeding, T/F: Answered incorrectly at Baseline and answered incorrectly at 3-Month Contact | 0
  Q15: See a doctor if you find unusual liquid coming from nipple when not pregnant/breastfeeding, T/F: Answered correctly at Baseline and answered incorrectly at 3-Month Contact | 2
  Q15: See a doctor if you find unusual liquid coming from nipple when not pregnant/breastfeeding, T/F: Answered correctly at Baseline and answered correctly at 3-Month Contact | 218
  Q16: See a doctor if you have a stabbing breast pain that does not seem to get better, T/F: Answered incorrectly at Baseline and answered correctly at 3-Month Contact | 4
  Q16: See a doctor if you have a stabbing breast pain that does not seem to get better, T/F: Answered incorrectly at Baseline and answered incorrectly at 3-Month Contact | 0
  Q16: See a doctor if you have a stabbing breast pain that does not seem to get better, T/F: Answered correctly at Baseline and answered incorrectly at 3-Month Contact | 1
  Q16: See a doctor if you have a stabbing breast pain that does not seem to get better, T/F: Answered correctly at Baseline and answered correctly at 3-Month Contact | 218
  Q17: See a doctor if you notice pulling in of the nipple or other parts of your breast(s), T/F: Answered incorrectly at Baseline and answered correctly at 3-Month Contact | 9
  Q17: See a doctor if you notice pulling in of the nipple or other parts of your breast(s), T/F: Answered incorrectly at Baseline and answered incorrectly at 3-Month Contact | 0
  Q17: See a doctor if you notice pulling in of the nipple or other parts of your breast(s), T/F: Answered correctly at Baseline and answered incorrectly at 3-Month Contact | 5
  Q17: See a doctor if you notice pulling in of the nipple or other parts of your breast(s), T/F: Answered correctly at Baseline and answered correctly at 3-Month Contact | 209
  Q18: Women don't need to be aware of changes with their breasts until they reach 40 years old, T/F: Answered incorrectly at Baseline and answered correctly at 3-Month Contact | 16
  Q18: Women don't need to be aware of changes with their breasts until they reach 40 years old, T/F: Answered incorrectly at Baseline and answered incorrectly at 3-Month Contact | 11
  Q18: Women don't need to be aware of changes with their breasts until they reach 40 years old, T/F: Answered correctly at Baseline and answered incorrectly at 3-Month Contact | 7
  Q18: Women don't need to be aware of changes with their breasts until they reach 40 years old, T/F: Answered correctly at Baseline and answered correctly at 3-Month Contact | 189
  Q19: Knowing how your breast/underarms normally look/feel are important parts of breast health, T/F: Answered incorrectly at Baseline and answered correctly at 3-Month Contact | 13
  Q19: Knowing how your breast/underarms normally look/feel are important parts of breast health, T/F: Answered incorrectly at Baseline and answered incorrectly at 3-Month Contact | 0
  Q19: Knowing how your breast/underarms normally look/feel are important parts of breast health, T/F: Answered correctly at Baseline and answered incorrectly at 3-Month Contact | 2
  Q19: Knowing how your breast/underarms normally look/feel are important parts of breast health, T/F: Answered correctly at Baseline and answered correctly at 3-Month Contact | 208
  Q20: A screening MAM is only needed if you noticed changes with your breast(s) in the past year, T/F: Answered incorrectly at Baseline and answered correctly at 3-Month Contact | 37
  Q20: A screening MAM is only needed if you noticed changes with your breast(s) in the past year, T/F: Answered incorrectly at Baseline and answered incorrectly at 3-Month Contact | 15
  Q20: A screening MAM is only needed if you noticed changes with your breast(s) in the past year, T/F: Answered correctly at Baseline and answered incorrectly at 3-Month Contact | 36
  Q20: A screening MAM is only needed if you noticed changes with your breast(s) in the past year, T/F: Answered correctly at Baseline and answered correctly at 3-Month Contact | 135
  Q21: When detected early, the chance of curing breast cancer is increased, T/F: Answered incorrectly at Baseline and answered correctly at 3-Month Contact | 2
  Q21: When detected early, the chance of curing breast cancer is increased, T/F: Answered incorrectly at Baseline and answered incorrectly at 3-Month Contact | 0
  Q21: When detected early, the chance of curing breast cancer is increased, T/F: Answered correctly at Baseline and answered incorrectly at 3-Month Contact | 4
  Q21: When detected early, the chance of curing breast cancer is increased, T/F: Answered correctly at Baseline and answered correctly at 3-Month Contact | 217
  Q22: Getting yearly MAM and clinical breast exams are the best ways to detect BC early, T/F: Answered incorrectly at Baseline and answered correctly at 3-Month Contact | 7
  Q22: Getting yearly MAM and clinical breast exams are the best ways to detect BC early, T/F: Answered incorrectly at Baseline and answered incorrectly at 3-Month Contact | 0
  Q22: Getting yearly MAM and clinical breast exams are the best ways to detect BC early, T/F: Answered correctly at Baseline and answered incorrectly at 3-Month Contact | 5
  Q22: Getting yearly MAM and clinical breast exams are the best ways to detect BC early, T/F: Answered correctly at Baseline and answered correctly at 3-Month Contact | 211
  Q23: BC is the most common cancer diagnosed among Hispanic/Latina women, T/F: Answered incorrectly at Baseline and answered correctly at 3-Month Contact | 42
  Q23: BC is the most common cancer diagnosed among Hispanic/Latina women, T/F: Answered incorrectly at Baseline and answered incorrectly at 3-Month Contact | 9
  Q23: BC is the most common cancer diagnosed among Hispanic/Latina women, T/F: Answered correctly at Baseline and answered incorrectly at 3-Month Contact | 14
  Q23: BC is the most common cancer diagnosed among Hispanic/Latina women, T/F: Answered correctly at Baseline and answered correctly at 3-Month Contact | 158
  Q24: Healthy women do not need to get MAM annually, T/F: Answered incorrectly at Baseline and answered correctly at 3-Month Contact | 25
  Q24: Healthy women do not need to get MAM annually, T/F: Answered incorrectly at Baseline and answered incorrectly at 3-Month Contact | 4
  Q24: Healthy women do not need to get MAM annually, T/F: Answered correctly at Baseline and answered incorrectly at 3-Month Contact | 11
  Q24: Healthy women do not need to get MAM annually, T/F: Answered correctly at Baseline and answered correctly at 3-Month Contact | 183
  Q25: If you don't see changes with your breasts in the past year, a MAM isn't necessary, T/F: Answered incorrectly at Baseline and answered correctly at 3-Month Contact | 39
  Q25: If you don't see changes with your breasts in the past year, a MAM isn't necessary, T/F: Answered incorrectly at Baseline and answered incorrectly at 3-Month Contact | 8
  Q25: If you don't see changes with your breasts in the past year, a MAM isn't necessary, T/F: Answered correctly at Baseline and answered incorrectly at 3-Month Contact | 9
  Q25: If you don't see changes with your breasts in the past year, a MAM isn't necessary, T/F: Answered correctly at Baseline and answered correctly at 3-Month Contact | 167
Statistical Analysis 1: Comparison: Living Room Visit Participants; Patients gave True/False responses to Question 1 at Baseline and 3-Month Contact; the True/False responses were mapped to being correct or incorrect. The null hypothesis was that the intervention had no effect on breast health, or that the probability of answering incorrectly on the Baseline questionnaire and correctly on the 3-Month Contact questionnaire was equal to the probability of answering correctly on the Baseline questionnaire and incorrectly on the 3-Month Contact questionnaire; Test type: Superiority; p = 0.2482, McNemar — Each of the 25 co-secondary objectives were tested at the 2-sided, Bonferroni-corrected alpha=0.002 significance level to preserve an overall type I error rate of 5%
Statistical Analysis 2: Comparison: Living Room Visit Participants; Patients gave True/False responses to Question 2 at Baseline and 3-Month Contact; the True/False responses were mapped to being correct or incorrect. The null hypothesis was that the intervention had no effect on breast health, or that the probability of answering incorrectly on the Baseline questionnaire and correctly on the 3-Month Contact questionnaire was equal to the probability of answering correctly on the Baseline questionnaire and incorrectly on the 3-Month Contact questionnaire; Test type: Superiority; p < .0001, McNemar — [p-value comment as in outcome 2, analysis 1]
Statistical Analysis 3: Comparison: Living Room Visit Participants; Patients gave True/False responses to Question 3 at Baseline and 3-Month Contact; the True/False responses were mapped to being correct or incorrect. The null hypothesis was that the intervention had no effect on breast health, or that the probability of answering incorrectly on the Baseline questionnaire and correctly on the 3-Month Contact questionnaire was equal to the probability of answering correctly on the Baseline questionnaire and incorrectly on the 3-Month Contact questionnaire; Test type: Superiority; p = 0.0050, McNemar — [p-value comment as in outcome 2, analysis 1]
Statistical Analysis 4: Comparison: Living Room Visit Participants; Patients gave True/False responses to Question 4 at Baseline and 3-Month Contact; the True/False responses were mapped to being correct or incorrect. The null hypothesis was that the intervention had no effect on breast health, or that the probability of answering incorrectly on the Baseline questionnaire and correctly on the 3-Month Contact questionnaire was equal to the probability of answering correctly on the Baseline questionnaire and incorrectly on the 3-Month Contact questionnaire; Test type: Superiority; p = 0.0423, McNemar — [p-value comment as in outcome 2, analysis 1]
Statistical Analysis 5: Comparison: Living Room Visit Participants; Patients gave True/False responses to Question 5 at Baseline and 3-Month Contact; the True/False responses were mapped to being correct or incorrect. The null hypothesis was that the intervention had no effect on breast health, or that the probability of answering incorrectly on the Baseline questionnaire and correctly on the 3-Month Contact questionnaire was equal to the probability of answering correctly on the Baseline questionnaire and incorrectly on the 3-Month Contact questionnaire; Test type: Superiority; p < .0001, McNemar — [p-value comment as in outcome 2, analysis 1]
Statistical Analysis 6: Comparison: Living Room Visit Participants; Patients gave True/False responses to Question 6 at Baseline and 3-Month Contact; the True/False responses were mapped to being correct or incorrect. The null hypothesis was that the intervention had no effect on breast health, or that the probability of answering incorrectly on the Baseline questionnaire and correctly on the 3-Month Contact questionnaire was equal to the probability of answering correctly on the Baseline questionnaire and incorrectly on the 3-Month Contact questionnaire; Test type: Superiority; p < .0001, McNemar — [p-value comment as in outcome 2, analysis 1]
Statistical Analysis 7: Comparison: Living Room Visit Participants; Patients gave True/False responses to Question 7 at Baseline and 3-Month Contact; the True/False responses were mapped to being correct or incorrect. The null hypothesis was that the intervention had no effect on breast health, or that the probability of answering incorrectly on the Baseline questionnaire and correctly on the 3-Month Contact questionnaire was equal to the probability of answering correctly on the Baseline questionnaire and incorrectly on the 3-Month Contact questionnaire; Test type: Superiority; p < .0001, McNemar — [p-value comment as in outcome 2, analysis 1]
Statistical Analysis 8: Comparison: Living Room Visit Participants; Patients gave True/False responses to Question 8 at Baseline and 3-Month Contact; the True/False responses were mapped to being correct or incorrect. The null hypothesis was that the intervention had no effect on breast health, or that the probability of answering incorrectly on the Baseline questionnaire and correctly on the 3-Month Contact questionnaire was equal to the probability of answering correctly on the Baseline questionnaire and incorrectly on the 3-Month Contact questionnaire; Test type: Superiority; p = 0.0002, McNemar — [p-value comment as in outcome 2, analysis 1]
Statistical Analysis 9: Comparison: Living Room Visit Participants; Patients gave True/False responses to Question 9 at Baseline and 3-Month Contact; the True/False responses were mapped to being correct or incorrect. The null hypothesis was that the intervention had no effect on breast health, or that the probability of answering incorrectly on the Baseline questionnaire and correctly on the 3-Month Contact questionnaire was equal to the probability of answering correctly on the Baseline questionnaire and incorrectly on the 3-Month Contact questionnaire; Test type: Superiority; p = 0.7456, McNemar — [p-value comment as in outcome 2, analysis 1]
Statistical Analysis 10: Comparison: Living Room Visit Participants; Patients gave True/False responses to Question 10 at Baseline and 3-Month Contact; the True/False responses were mapped to being correct or incorrect. The null hypothesis was that the intervention had no effect on breast health, or that the probability of answering incorrectly on the Baseline questionnaire and correctly on the 3-Month Contact questionnaire was equal to the probability of answering correctly on the Baseline questionnaire and incorrectly on the 3-Month Contact questionnaire; Test type: Superiority; p < .0001, McNemar — [p-value comment as in outcome 2, analysis 1]
Statistical Analysis 11: Comparison: Living Room Visit Participants; Patients gave True/False responses to Question 11 at Baseline and 3-Month Contact; the True/False responses were mapped to being correct or incorrect. The null hypothesis was that the intervention had no effect on breast health, or that the probability of answering incorrectly on the Baseline questionnaire and correctly on the 3-Month Contact questionnaire was equal to the probability of answering correctly on the Baseline questionnaire and incorrectly on the 3-Month Contact questionnaire; Test type: Superiority; p = 0.0028, McNemar — [p-value comment as in outcome 2, analysis 1]
Statistical Analysis 12: Comparison: Living Room Visit Participants; Patients gave True/False responses to Question 12 at Baseline and 3-Month Contact; the True/False responses were mapped to being correct or incorrect. The null hypothesis was that the intervention had no effect on breast health, or that the probability of answering incorrectly on the Baseline questionnaire and correctly on the 3-Month Contact questionnaire was equal to the probability of answering correctly on the Baseline questionnaire and incorrectly on the 3-Month Contact questionnaire; Test type: Superiority; p = 0.0707, McNemar — [p-value comment as in outcome 2, analysis 1]
Statistical Analysis 13: Comparison: Living Room Visit Participants; Patients gave True/False responses to Question 13 at Baseline and 3-Month Contact; the True/False responses were mapped to being correct or incorrect. The null hypothesis was that the intervention had no effect on breast health, or that the probability of answering incorrectly on the Baseline questionnaire and correctly on the 3-Month Contact questionnaire was equal to the probability of answering correctly on the Baseline questionnaire and incorrectly on the 3-Month Contact questionnaire; Test type: Superiority; p = 0.0026, McNemar — [p-value comment as in outcome 2, analysis 1]
Statistical Analysis 14: Comparison: Living Room Visit Participants; Patients gave True/False responses to Question 14 at Baseline and 3-Month Contact; the True/False responses were mapped to being correct or incorrect. The null hypothesis was that the intervention had no effect on breast health, or that the probability of answering incorrectly on the Baseline questionnaire and correctly on the 3-Month Contact questionnaire was equal to the probability of answering correctly on the Baseline questionnaire and incorrectly on the 3-Month Contact questionnaire; Test type: Superiority; p = 0.1797, McNemar — [p-value comment as in outcome 2, analysis 1]
Statistical Analysis 15: Comparison: Living Room Visit Participants; Patients gave True/False responses to Question 15 at Baseline and 3-Month Contact; the True/False responses were mapped to being correct or incorrect. The null hypothesis was that the intervention had no effect on breast health, or that the probability of answering incorrectly on the Baseline questionnaire and correctly on the 3-Month Contact questionnaire was equal to the probability of answering correctly on the Baseline questionnaire and incorrectly on the 3-Month Contact questionnaire; Test type: Superiority; p = 0.6547, McNemar — [p-value comment as in outcome 2, analysis 1]
Statistical Analysis 16: Comparison: Living Room Visit Participants; Patients gave True/False responses to Question 16 at Baseline and 3-Month Contact; the True/False responses were mapped to being correct or incorrect. The null hypothesis was that the intervention had no effect on breast health, or that the probability of answering incorrectly on the Baseline questionnaire and correctly on the 3-Month Contact questionnaire was equal to the probability of answering correctly on the Baseline questionnaire and incorrectly on the 3-Month Contact questionnaire; Test type: Superiority; p = 0.1797, McNemar — [p-value comment as in outcome 2, analysis 1]
Statistical Analysis 17: Comparison: Living Room Visit Participants; Patients gave True/False responses to Question 17 at Baseline and 3-Month Contact; the True/False responses were mapped to being correct or incorrect. The null hypothesis was that the intervention had no effect on breast health, or that the probability of answering incorrectly on the Baseline questionnaire and correctly on the 3-Month Contact questionnaire was equal to the probability of answering correctly on the Baseline questionnaire and incorrectly on the 3-Month Contact questionnaire; Test type: Superiority; p = 0.2850, McNemar — [p-value comment as in outcome 2, analysis 1]
Statistical Analysis 18: Comparison: Living Room Visit Participants; Patients gave True/False responses to Question 18 at Baseline and 3-Month Contact; the True/False responses were mapped to being correct or incorrect. The null hypothesis was that the intervention had no effect on breast health, or that the probability of answering incorrectly on the Baseline questionnaire and correctly on the 3-Month Contact questionnaire was equal to the probability of answering correctly on the Baseline questionnaire and incorrectly on the 3-Month Contact questionnaire; Test type: Superiority; p = 0.0606, McNemar — [p-value comment as in outcome 2, analysis 1]
Statistical Analysis 19: Comparison: Living Room Visit Participants; Patients gave True/False responses to Question 19 at Baseline and 3-Month Contact; the True/False responses were mapped to being correct or incorrect. The null hypothesis was that the intervention had no effect on breast health, or that the probability of answering incorrectly on the Baseline questionnaire and correctly on the 3-Month Contact questionnaire was equal to the probability of answering correctly on the Baseline questionnaire and incorrectly on the 3-Month Contact questionnaire; Test type: Superiority; p = 0.0045, McNemar — [p-value comment as in outcome 2, analysis 1]
Statistical Analysis 20: Comparison: Living Room Visit Participants; Patients gave True/False responses to Question 20 at Baseline and 3-Month Contact; the True/False responses were mapped to being correct or incorrect. The null hypothesis was that the intervention had no effect on breast health, or that the probability of answering incorrectly on the Baseline questionnaire and correctly on the 3-Month Contact questionnaire was equal to the probability of answering correctly on the Baseline questionnaire and incorrectly on the 3-Month Contact questionnaire; Test type: Superiority; p = 0.9068, McNemar — [p-value comment as in outcome 2, analysis 1]
Statistical Analysis 21: Comparison: Living Room Visit Participants; Patients gave True/False responses to Question 21 at Baseline and 3-Month Contact; the True/False responses were mapped to being correct or incorrect. The null hypothesis was that the intervention had no effect on breast health, or that the probability of answering incorrectly on the Baseline questionnaire and correctly on the 3-Month Contact questionnaire was equal to the probability of answering correctly on the Baseline questionnaire and incorrectly on the 3-Month Contact questionnaire; Test type: Superiority; p = 0.4142, McNemar — [p-value comment as in outcome 2, analysis 1]
Statistical Analysis 22: Comparison: Living Room Visit Participants; Patients gave True/False responses to Question 22 at Baseline and 3-Month Contact; the True/False responses were mapped to being correct or incorrect. The null hypothesis was that the intervention had no effect on breast health, or that the probability of answering incorrectly on the Baseline questionnaire and correctly on the 3-Month Contact questionnaire was equal to the probability of answering correctly on the Baseline questionnaire and incorrectly on the 3-Month Contact questionnaire; Test type: Superiority; p = 0.5637, McNemar — [p-value comment as in outcome 2, analysis 1]
Statistical Analysis 23: Comparison: Living Room Visit Participants; Patients gave True/False responses to Question 23 at Baseline and 3-Month Contact; the True/False responses were mapped to being correct or incorrect. The null hypothesis was that the intervention had no effect on breast health, or that the probability of answering incorrectly on the Baseline questionnaire and correctly on the 3-Month Contact questionnaire was equal to the probability of answering correctly on the Baseline questionnaire and incorrectly on the 3-Month Contact questionnaire; Test type: Superiority; p = 0.0002, McNemar — [p-value comment as in outcome 2, analysis 1]
Statistical Analysis 24: Comparison: Living Room Visit Participants; Patients gave True/False responses to Question 24 at Baseline and 3-Month Contact; the True/False responses were mapped to being correct or incorrect. The null hypothesis was that the intervention had no effect on breast health, or that the probability of answering incorrectly on the Baseline questionnaire and correctly on the 3-Month Contact questionnaire was equal to the probability of answering correctly on the Baseline questionnaire and incorrectly on the 3-Month Contact questionnaire; Test type: Superiority; p = 0.0196, McNemar — [p-value comment as in outcome 2, analysis 1]
Statistical Analysis 25: Comparison: Living Room Visit Participants; Patients gave True/False responses to Question 25 at Baseline and 3-Month Contact; the True/False responses were mapped to being correct or incorrect. The null hypothesis was that the intervention had no effect on breast health, or that the probability of answering incorrectly on the Baseline questionnaire and correctly on the 3-Month Contact questionnaire was equal to the probability of answering correctly on the Baseline questionnaire and incorrectly on the 3-Month Contact questionnaire; Test type: Superiority; p < .0001, McNemar — This outcome measure for Q25 was tested at the 2-sided, Bonferroni-corrected alpha=0.002 significance level to preserve an overall type I error rate of 5% in the analyses of 25 questions

ADVERSE EVENTS:
Time Frame: Adverse events were not collected for the study as the breast health education program was unlikely to present harm to the subjects enrolled in this study.
Description: The number of participants at risk for All-Cause Mortality is zero because adverse events were not monitored/assessed.
  The number of participants at risk for Serious Adverse Events is zero because adverse events were not monitored/assessed.
  The number of participants at risk for Other (Not Including Serious) Adverse Events is zero because adverse events were not monitored/assessed.
Arm/Group | Living Room Visit Participants
All-Cause Mortality (participants affected / at risk) | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

LIMITATIONS AND CAVEATS:
Roughly 32% (32.22%) of patients were non-compliant in returning three-month phone call (due to changed contact information or study team attempted three phone call contacts as defined in protocol).

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes